CLINICAL TRIAL: NCT05311592
Title: Montefiore Medical Center Supporting Responsible Fatherhood Program
Brief Title: Supporting Responsible Fatherhood Program (Fatherhood FIRE)
Acronym: FIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); BronxWorks (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-12757
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Parenting; Family Relations; Father-Child Relations

STUDY DESIGN:
Intervention Model Description: The investigator will run workshops virtually, through Zoom, and in person. Participants will be randomized either to the virtual condition, or to the in person condition.
  Update: Effective 1/1/2025 randomization ceased and from that date onward data participants were able to choose which arm they partook in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In Person (Experimental): Participants will receive all services in person, including participating in the initial intake process, and attending all workshops.
  Interventions: Behavioral: HERO Dads Program
- Virtual (Zoom) (Experimental): Participants will complete their intake process in person, but will complete all workshops virtually through Zoom.
  Interventions: Behavioral: HERO Dads Program

INTERVENTIONS:
Behavioral: HERO Dads Program — The HERO Dads Program is a 4-week series of workshops for non-custodial fathers that focuses on improving parenting, offering job support, and financial counseling.

SUMMARY:
Montefiore Medical Center (in partnership with BronxWorks) is implementing a large-scope program to promote responsible fatherhood in the Bronx among low-income adult (18 years or older) fathers with non-custodial children (under the age of 24). The program, called HERO Dads (Healthy, Empowered, Resilient, Open Dads), will promote responsible fatherhood by enhancing relationship and anger-management skills and providing marriage education; providing skills-based parenting education, disseminating information about good parenting practices, and encouraging child support payments (in partnership with our local OCSE); and fostering economic stability by providing employment-related supports inclusive of job search, vocational skills training, job referrals, and job retention.

DETAILED DESCRIPTION:
The program model is based on the premise that relationship and parenting skills can be taught, and will lead to improvements in relationships (knowledge about relationships, communication skills, stress management, reduction in destructive conflict), parenting (knowledge about child development, engagement with non-custodial children, effective parenting, co-parent communication, child well-being), and economic status (vocational skills, new employment or career advancement, financial literacy, child support). The investigator will provide core relationship and relationship education workshops using an empirically supported curriculum (24/7 Dad) plus employment workshops, numerous supplemental activities to promote responsible fatherhood, individualized vocational case management, and job-driven employment services. In total, the investigator expects to enroll 1,475 non-custodial fathers in the program and provide an average of 34 hours of total programming per participant (including 24 hours of core workshops), which the investigator believes is a sufficient dosage to detect impacts.

ELIGIBILITY:
Inclusion Criteria:

* Non-custodial fathers who are 18 years or older
* Have non-custodial children (biological, foster, adopted) under the age of 24
* Income below 200% poverty line

Exclusion Criteria:

* Active intimate partner violence and increased risk of intimate partner violence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Fatherhood Involvement | Change from Baseline to 6 months after intervention
  Fatherhood Involvement will be assessed using the Inventory of Fatherhood Involvement short form (IFI) questionnaire. The IFI is a 26-item self-report instrument that assesses indirect and direct father involvement using a 7- point Likert scale ranging from 0 (very poor) to 6 (excellent). This measure addresses the 3 main domains of father involvement: engagement, accessibility, and responsibility. Overall scores can therefore range from 0 to 156. Higher scores represent increased levels of engagement. Scores will be summarized by study arm using basic descriptive statistics. 2-sample t-test will be used to compare the changes in the IFI scores from Baseline to 6-month follow-up between the study arms.

SECONDARY OUTCOMES:
Emotional Intelligence | Baseline
  Emotional Intelligence will be assessed using the Assessing Emotions Scale. The Assessing Emotions Scale is a 33-item self-report inventory focusing on typical emotional intelligence. Participants provide responses using a 5-item Likert scale of measurement with values ranging from 1 ("strongly disagree") to 5 ("strongly agree"). Total scale scores are calculated by reverse coding items 5, 28, and 33 and then summing the responses across all items. The overall scoring range is 33-166, with higher scores indicating more characteristic emotional intelligence. Scores will be summarized by study arm using basic descriptive statistics.
Quality of Co-Parenting Relationships | Baseline
  Quality of Co-Parenting Relationships will be evaluated using the Parenting Alliance Inventory (PAI). The PAI is a 20 item self-report instrument that assesses the degree to which parents believe that they have a sound working relationship with their child's other parent. Participants provide responses to the PAI using a 5-point Likert scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), yielding an overall possible score of 20-100. Higher PAI scores are indicative of a stronger, more positive parenting alliance. Results will be summarized by study arm using basic descriptive statistics.
Parent-Child Relationship Quality | Baseline
  Parent-Child Relationship Quality will be assessed using the Child-Parent Relationship Scale Short Form (CPRS-SF). The CPRS-SF is a 15-item self-report measure that assesses parents' perceptions of their relationship with their child, especially related to closeness and conflict. Items are rated on a 5-point scale ranging from 1 ("Definitely does not apply") to 5 ("Definitively applies"). Items 2, 4, 8, 10, 11, 12, 13, 14 comprise the Conflict subscale and measure the degree to which a parent feels that his or her relationship with a child is characterized by negativity. Items 1, 3, 5, 6, 7, 9, 15 comprise the Closeness subscale and measure the extent to which a parent feels that the relationship is characterized by warmth, affection, and open communication. Higher scores for each subscale are indicative of more Conflict or Closeness, respectively. A composite score is obtained by summing item responses for each subscale, yielding an overall possible scoring range of 15-75.
Skills/Knowledge Assessment (Skills/Knowledge Acquisition) | Change from Baseline to 6 months after intervention
  The Skills/Knowledge Assessment is an outcome measure that will be developed by program staff together with the local evaluator. This 14-item measure is a multiple-choice assessment using scenarios describing parent-child and co-parenting interactions to determine whether fathers have learned skills and techniques taught at workshops. This measure will be calculated by obtaining the percentage of correctly scored items. Higher scores indicate greater skill acquisition. Two versions of this assessment will be created to prevent practice effects. Given that this is a homegrown measure, to validate this measure the investigators will correlate the skill assessment scores with the Assessing Emotions Scale and assess whether relationship skill scores differ by key demographic and social economic factors. Results will be summarized by study arm using basic descriptive statistics.
Childhood Trauma | Baseline
  Childhood Trauma will be assessed using the Childhood Trauma Questionnaire Short Form (CTQ-SF). The CTQ-SF is a 25-item measure of childhood trauma covering 5 trauma types: Emotional/Physical/Sexual Abuse, Emotional Neglect and Physical Neglect along with a separate Minimization/Denial scale. Participants respond to each item using a 5-point Likert scale ranging from 1 ("Never true") to 5 ("Very often true"), yielding an overall possible score of 25-125 such that higher scores are indicative of increased childhood trauma. Seven of the items must be reverse-coded (i.e., 1=5, 2=4, 3=3, 4=2, 5=1) before summing. Results will be summarized by study arm using basic descriptive statistics.

OTHER OUTCOMES:
Information, Family Outcomes, Reporting, and Management (nFORM) Applicant Characteristics | Baseline
  This is a survey developed by the Office of Family Assistance utilized by all grantees participating in the national study, that gathers demographic information regarding participants.
Information, Family Outcomes, Reporting, and Management (nFORM) Pre-Program Survey | At start of intervention (Week 1 of 4)
  This is a survey developed by the Office of Family Assistance utilized by all grantees participating in the national study that includes questions regarding relationship satisfaction, financial stability, and parenting.
Information, Family Outcomes, Reporting, and Management (nFORM) Post-Program Survey | Immediately post intervention (Week 4 of 4 weeks)
  This is a survey developed by the Office of Family Assistance utilized by all grantees participating in the national study that includes questions regarding relationship satisfaction, financial stability, and parenting.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wetzler, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawkins, A. (2019) Are federally-supported relationship education programs for lower-income individuals and couples working? A review of evaluation research. American Enterprise Institute.
- [Background] Haskins, R. & Sawhill, I. (2003) Work and marriage: The way to end poverty and welfare. The Brookings Institution Policy Brief: Welfare Reform and Beyond #28, 1-8.
- [Background] Acs, G. & Nelson, S. (2004) What do 'I do's do? Potential benefits of marriage for cohabiting couples with children." Assessing the New Federalism Policy Brief B-59. Washington, DC: The Urban Institute.
- [Background] Kiecolt-Glaser JK, Newton TL. Marriage and health: his and hers. Psychol Bull. 2001 Jul;127(4):472-503. doi: 10.1037/0033-2909.127.4.472. PMID 11439708
- [Background] Bramlett MD, Mosher WD. Cohabitation, marriage, divorce, and remarriage in the United States. Vital Health Stat 23. 2002 Jul;(22):1-93. PMID 12183886
- [Background] McLanahan, S., Garfinkel, I., Reichman, N. et al. (2003) The Fragile Families and Child Wellbeing Study: Baseline National Report. Princeton, NJ: Center for Research on Child Wellbeing, Princeton University.
- [Background] Carlson MJ, McLanahan SS, Brooks-Gunn J. Coparenting and nonresident fathers' involvement with young children after a nonmarital birth. Demography. 2008 May;45(2):461-88. doi: 10.1353/dem.0.0007. PMID 18613490
- [Background] Carlson MJ, VanOrman AG, Turner KJ. Fathers' Investments of Money and Time Across Residential Contexts. J Marriage Fam. 2017 Feb;79(1):10-23. doi: 10.1111/jomf.12324. Epub 2016 Jun 27. PMID 29681652
- [Background] Amato, P. R. (2000). Consequences of divorce for adults and children. Journal of Marriage and Family, 58, 356 365.
- [Background] Amato PR. Children of divorce in the 1990s: an update of the Amato and Keith (1991) meta-analysis. J Fam Psychol. 2001 Sep;15(3):355-70. doi: 10.1037//0893-3200.15.3.355. PMID 11584788
- [Background] Amato PR, Booth A. The legacy of parents' marital discord: consequences for children's marital quality. J Pers Soc Psychol. 2001 Oct;81(4):627-38. PMID 11642350
- [Background] Whisman, M. A., & Uebelacker, L. A. (2003). Comorbidity of relationship distress and mental and physical health problems. In D. K. Snyder & M. A. Whisman (Eds.), Treating difficult couples (pp. 3-26). New York, NY: Guilford.
- [Background] Institute for American Values (2002). Why marriage matters: Twenty-one conclusions from the social sciences.
- [Background] Yoder, J., Brisson, D. & Lopez, A. (2016) Moving beyond fatherhood involvement: The association between father-child relationship quality and youth delinquency trajectories. Family Relations, 65: 462-476.
- [Background] Cabrera, N. & Tamis-LeMonda, C. (Eds.) (2013) Handbook of Father Involvement: Multidisciplinary Perspectives (2nd Ed). New York, NY: Routledge
- [Background] Hawkins, A. J., & Fackrell, T. A. (2010). Does couple education for lower-income couples work? A meta-analytic study of emerging research. Journal of Couple & Relationship Therapy: Innovations in Clinical and Educational Interventions, 9(2), 181-191.
- [Background] Cummings, E. & Merrilees, C. (2010) Identifying the dynamic processes underlying links between marital conflict and child adjustment. In M. Schulz, M. Pruett, P. Kerig & R. Parke (Eds.) Strengthening couple relationships for optimal child development: Lessons from research and intervention (pp. 27-40). Washington, D.C.: American Psychological Association.
- [Background] Gottman,J.M., Coan, J. A., Carrere, S., & Swanson, C. (1998). Predicting marital happiness and stability from newlywed interactions. Journal of Marriage and Family, 60, 5-22.
- [Background] Markman, H. J., & Hahlweg, K. (1993). The prediction & prevention of marital distress: An international perspective. Clinical Psychology Review, 13, 29-43.
- [Background] Gottman, J. M. (1994). What predicts divorce? The relationship between marital processes and marital outcomes. Hillsdale, NJ: Erlbaum.
- [Background] Wetzler, S. Government-funded relationship education can work, The Atlantic, March 14, 2014.
- [Background] Hsueh, J., Alderson, D. P., Lundquist, E., Michalopoulos, C., Gubits, D., Fein, D., & Knox, V. (2012). The Supporting Healthy Marriage evaluation: Early impacts on low-income families (OPRE Report No. 2012-11). Washington, DC: U.S. Department of Health and Human Services, Administration for Children and Families, Office of Planning, Research and Evaluation.
- [Background] Lundquist, E., Hsueh, J., Lowenstein, A., Faucetta, K., Gubits, D., Michalopoulos, C., & Knox, V. (2014). A family strengthening program for low-income families: Final impacts from the Supporting Healthy Marriage evaluation. OPRE Report 2013-49A. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U. S. Department of Health and Human Services.
- [Background] Cowan, P. & Cowan, C. (2014). Controversies in couple relationship education: Overlooked evidence and implications for research and policy. Psychology, Public Policy, and Law, 20, 361-383.
- [Background] Hawkins AJ, Blanchard VL, Baldwin SA, Fawcett EB. Does marriage and relationship education work? A meta-analytic study. J Consult Clin Psychol. 2008 Oct;76(5):723-34. doi: 10.1037/a0012584. PMID 18837590
- [Background] Hawkins AJ, Stanley SM, Blanchard VL, Albright M. Exploring programmatic moderators of the effectiveness of marriage and relationship education programs: a meta-analytic study. Behav Ther. 2012 Mar;43(1):77-87. doi: 10.1016/j.beth.2010.12.006. Epub 2011 Jun 1. PMID 22304880
- [Background] Pinquart, M., & Teubert, D. (2010). A meta-analytic study of couple interventions during the transition to parenthood. Family Relations, 59, 221-231.
- [Background] Wood, R., McConnell, S., Quinn, M., Clarkwest, A., & Hsueh, J. (2010). Strengthening Unmarried parents' relationships: The early impacts of building strong families. Washington DC: Mathematic Policy Research.
- [Background] Schutte, N. S., Malouff, J. M., Hall, L. E., Haggerty, D. J., Cooper, J. T., Golden, C. J., & Dornheim, L. (1998). Development and validation of a measure of emotional intelligence. Personality and Individual Differences, 25(2), 167-177.
- [Background] Abidin, R. R., & Brunner, J. F. (1995). Development of a parenting alliance inventory. Journal of Clinical Child Psychology, 24(1), 31-40.
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Driscoll, K., & Pianta, R. C. (2011). Mothers' and fathers' perceptions of conflict and closeness in parent-child relationships during early childhood. Journal of Early Childhood & Infant Psychology, (7).
- [Background] Hawkins, A. J., Bradford, K. P., Palkovitz, R., Christiansen, S. L., Day, R. D., & Call, V. R. (2002). The inventory of father involvement: A pilot study of a new measure of father involvement. The Journal of Men's Studies, 10(2), 183-196.
- [Background] Lamb, M. E., Pleck, J. H., Charnov, E. L., & Levine, J. A. (1987). A biosocial perspective on paternal behavior and involvement. In J. B. Lancaster, J. Altmann, A. S. Rossi, & L. R. Sherrod (Eds.), Parenting across the lifespan: Biosocial perspectives (pp. 111-142). Hawthorne, NY: Aldine.
- See also: Married and poor: Basic characteristics of economically disadvantaged married couples in the US. Working Paper SHM-01, Supporting Healthy Marriage Project, New York: MDRC — http://www.mdrc.org/publications/393/workpaper.html
- See also: Implementing an innovative parenting program for fathers: Findings from the B3 study OPRE Report 2019-111. — https://www.mdrc.org/sites/default/files/innovative_parenting_b3_findings_dec_2019_0.pdf

DOCUMENTS (1):
  • Informed Consent Form (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT05311592/ICF_000.pdf